CLINICAL TRIAL: NCT05353751
Title: Examining the Effectiveness of a Mindfulness-based Intervention for Underserved Adolescents With and Without Caregiver Involvement
Brief Title: Kind Minds Program for Youth With Anxiety and Depression
Acronym: KMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Denise A. Chavira, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-001218
Record Dates: First submitted 2022-02-02; First posted 2022-04-29 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Child Anxiety; Depression
Keywords: mindfulness; children; adolescents; anxiety; depression
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kind Minds Program -Family (Experimental): In the Family condition (KMP-Fam), both caregiver and adolescent will receive the KMP intervention via an online mindfulness program, augmented by weekly video conference support from a Community Health Worker (CHW) Kindness Coach
  Interventions: Behavioral: Kind Minds Program
- Kind Minds Program -Teen Only (Active Comparator): In the Teen-Only condition (KMP-TO), only the adolescent will receive the KMP intervention via an online mindfulness program augmented by weekly video conference support from a CHW Kindness Coach.
  Interventions: Behavioral: Kind Minds Program

INTERVENTIONS:
Behavioral: Kind Minds Program — The KMP intervention uses an online mindfulness phone based program. During the 9-week program, Community Health Worker (CHW) Kindness Coaches will meet weekly for 30 minutes via Zoom with either a) the caregiver and adolescent (in separate meetings), or b) the adolescent only to review and complete a new "session" using the online mindfulness program. Participants will be prompted to complete mindfulness activities between sessions by notifications, conducive to their school and work schedules. Weekly content and meditations/activities focus on mindfulness skills of present moment awareness, nonjudgment, compassion, and gratitude.

SUMMARY:
Rates of anxiety and depression in youth are substantial, causing a major unmet need for effective interventions. Participation in mindfulness interventions has been demonstrated to reduce anxiety and depressive symptoms among teenagers. Parents' participation in mindfulness interventions has also been shown to reduce their children's mental health symptoms. However, there is no available evidence regarding potential additional benefits for adolescents' mental health of having both the adolescent and their parent or caregiver learn and practice mindfulness simultaneously.

This pilot intervention study aims to explore potential additive effects of parent/caregiver participation in a digitally-based, kindness-focused, coached mindfulness intervention program for adolescents that lasts 9 weeks. Participating parent/caregiver-child pairs (n = 30) will include one teenager between 12 and 17 years old with a current diagnosis of an anxiety or depressive disorder and one parent/caregiver. All adolescent participants will take part in the mindfulness intervention. Half of the parents/caregivers will be randomized to also take part in the mindfulness program. Outcomes will be compared between families in which only the teen participates in the mindfulness program and families in which the teen and parent/caregiver participate in the intervention.

Adolescents and parents/caregivers will take part in evaluations before, in the middle of, and after the end of the mindfulness program, meaning that participation in the study will take a total of approximately 12 weeks. Pre, mid, and post evaluations will include online questionnaires. Pre and post evaluations will also include clinical interviews via phone or video conference. Evaluations will include measures of mental health diagnoses and symptoms, mood, interpersonal and family functioning, mindfulness, and perceptions of/satisfaction with the program. Participating adolescents and parents/caregivers will also fill out weekly brief questionnaires of anxiety and depressive symptoms. The primary outcome of interest is adolescent mental health, including anxiety and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include:

  1. one adolescent (aged 12-17 years) with a current diagnosis of an anxiety or depressive disorder)
  2. one of their parents/caregivers.
  3. Both adolescent and caregiver must speak English to the degree necessary to participate in the intervention program, which is only available in English.
  4. Parent and youth must have a smart phone and be willing to download the online mindfulness program.

Exclusion Criteria:

* Exclusion criteria apply to both caregiver and adolescent and include:

  1. current alcohol or substance use disorder or suicidality
  2. lifetime diagnosis of bipolar disorder, schizophrenia, autism, conduct disorder, or developmental delay diagnosed by an independent evaluator;
  3. English reading level below 4th grade
  4. non English speaking
  5. currently receiving mindfulness-based mental health services or taking medication to treat anxiety or depression.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | 12-14 weeks after baseline assessment
  self report of depressive symptoms
Generalized Anxiety Disorder-7 | 12-14 weeks after baseline assessment
  self report of anxiety symptoms
SCARED -Screen for child anxiety and related emotional disorders | 12-14 weeks after baseline assessment
  self report of anxiety symptoms

SECONDARY OUTCOMES:
Kiddie Schedule for Affective Disorders and Schizophrenia interview -anxiety and depressive disorder modules | 12-14 weeks after baseline assessment
  remission on primary anxiety or primary depressive disorder diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Chavira, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Imperial High School, Imperial, California, United States

IPD SHARING:
Plan to Share IPD: No